CLINICAL TRIAL: NCT03806114
Title: Impact of Dislocation Precautions on Fear and Function in Patients Undergoing Hip Replacement
Brief Title: Dislocation Precautions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20180880
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Arthroplasty, Hip Replacement; Arthroplasties, Hip Replacement; Health-Related Quality Of Life

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Anterior Approach Precautions (Other): This group receives precautions and have a total hip arthroplasty with a posterior approach.
  Interventions: Procedure: Anterior Approach Precautions
- Posterior Approach Precautions (Other): This group receives precautions and have a total hip arthroplasty with a posterior approach.
  Interventions: Procedure: Posterior Approach Precautions
- Anterior Approach No Precautions (Other): This group receives does not precautions and have a total hip arthroplasty with an anterior approach.
  Interventions: Procedure: No Precautions
- Posterior Approach No Precautions (Other): This group receives does not receive precautions and have a total hip arthroplasty with a posterior approach.
  Interventions: Procedure: No Precautions

INTERVENTIONS:
Procedure: Posterior Approach Precautions — These patients will be advised not to bend their leg or trunk more than 90 degrees, avoid crossing the leg or crossing midline, and rotating the leg inwards. Patients will also be instructed to put a pillow in between their legs while sleeping for 6 weeks and to avoid bathing for 6 weeks.
  Arms: Posterior Approach Precautions
Procedure: Anterior Approach Precautions — These patients will be advised to avoid extending the leg back, rotating the leg outwards, and lifting their bottom when lying down after their surgery for 6 weeks.
  Arms: Anterior Approach Precautions
Procedure: No Precautions — For the non-precautions group, there will be no mention of precautions by any providers before, during, and after surgery. No equipment will be given, but a list of self-care equipment will be available for 'comfort' purposes. Patients will be instructed to avoid bathing for 4 weeks. All groups will have instructions to use a walking aid and a toilet seat if needed, to weight-bear as tolerated, and to avoid driving for 3 weeks.
  Arms: Anterior Approach No Precautions; Posterior Approach No Precautions

SUMMARY:
This study is looking at the impact of giving patients precautions, or restrictions for movement, when undergoing a total hip replacement. Have of the participants will receive precautions, while the other half will not receive any precautions.

DETAILED DESCRIPTION:
Patients undergoing hip replacements are often told by health care providers to avoid specific positions and activities to decrease the risk of their hip dislocating following their surgery. This, however, results in patients becoming more fearful of moving and leads to limitations in their function and decreased quality of life. Previous research has shown that hip dislocations following surgery are most commonly attributed to poor implant position rather than the actions of the patients. Teaching precautions takes up healthcare resources and may use finances that are not necessarily required. This study aims to compare groups with half receiving precautions and half not receiving precautions, to assess the impact of precautions on the patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Receiving a primary total hip arthroplasty (THA) due to osteoarthritis or osteonecrosis
* Over 18
* Willing and able to sign consent

Exclusion Criteria:

* Receiving a lateral approach hip arthroplasty
* Cannot make follow up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2023-06-21 (Estimated); Study Completion 2023-12-21 (Estimated)

PRIMARY OUTCOMES:
Change in Oxford Hip Score | Week before surgery to 6 months after surgery
  Assess function of the hip

SECONDARY OUTCOMES:
Change in Tampa Scale for Kinesiophobia | Week before surgery to 6 months after surgery
  This assesses kinesiophobia, using a 17 item scale with each item using a 4 point Likert scale . The final score is the sum of all questions except for 4, 8, 12 and 16 which has their score inverted before being added. The final score ranges from from 17-68 points with 68 being the highest degree of kinesiophobia.
Change in Forgotten Joint Score | 6 weeks after surgery to 6 months after surgery
  This measures awareness of a replaced joint
Change in EQ-5D-5L | Week before surgery to 6 months after surgery
  This measures general health
Canadian Patient Experience Survey - Inpatient Care (CPES-IC) | At 2 weeks after surgery
  This will measure the patients' experience.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Seagrave KG, Troelsen A, Malchau H, Husted H, Gromov K. Acetabular cup position and risk of dislocation in primary total hip arthroplasty. Acta Orthop. 2017 Feb;88(1):10-17. doi: 10.1080/17453674.2016.1251255. Epub 2016 Nov 23. PMID 27879150
- [Background] Smith TO, Jepson P, Beswick A, Sands G, Drummond A, Davis ET, Sackley CM. Assistive devices, hip precautions, environmental modifications and training to prevent dislocation and improve function after hip arthroplasty. Cochrane Database Syst Rev. 2016 Jul 4;7(7):CD010815. doi: 10.1002/14651858.CD010815.pub2. PMID 27374001
- [Background] van der Weegen W, Kornuijt A, Das D. Do lifestyle restrictions and precautions prevent dislocation after total hip arthroplasty? A systematic review and meta-analysis of the literature. Clin Rehabil. 2016 Apr;30(4):329-39. doi: 10.1177/0269215515579421. Epub 2015 Mar 31. PMID 25834275
- [Background] Barnsley L, Barnsley L, Page R. Are Hip Precautions Necessary Post Total Hip Arthroplasty? A Systematic Review. Geriatr Orthop Surg Rehabil. 2015 Sep;6(3):230-5. doi: 10.1177/2151458515584640. PMID 26328242
- [Background] Westby MD, Brittain A, Backman CL. Expert consensus on best practices for post-acute rehabilitation after total hip and knee arthroplasty: a Canada and United States Delphi study. Arthritis Care Res (Hoboken). 2014 Mar;66(3):411-23. doi: 10.1002/acr.22164. PMID 24023047
- [Background] Vissers MM, Bussmann JB, Verhaar JA, Busschbach JJ, Bierma-Zeinstra SM, Reijman M. Psychological factors affecting the outcome of total hip and knee arthroplasty: a systematic review. Semin Arthritis Rheum. 2012 Feb;41(4):576-88. doi: 10.1016/j.semarthrit.2011.07.003. Epub 2011 Oct 28. PMID 22035624
- [Background] Swinkels-Meewisse EJ, Swinkels RA, Verbeek AL, Vlaeyen JW, Oostendorp RA. Psychometric properties of the Tampa Scale for kinesiophobia and the fear-avoidance beliefs questionnaire in acute low back pain. Man Ther. 2003 Feb;8(1):29-36. doi: 10.1054/math.2002.0484. PMID 12586559
- [Background] Pincus T, Vogel S, Burton AK, Santos R, Field AP. Fear avoidance and prognosis in back pain: a systematic review and synthesis of current evidence. Arthritis Rheum. 2006 Dec;54(12):3999-4010. doi: 10.1002/art.22273. PMID 17133530
- [Background] Darlow B, Fullen BM, Dean S, Hurley DA, Baxter GD, Dowell A. The association between health care professional attitudes and beliefs and the attitudes and beliefs, clinical management, and outcomes of patients with low back pain: a systematic review. Eur J Pain. 2012 Jan;16(1):3-17. doi: 10.1016/j.ejpain.2011.06.006. PMID 21719329
- [Background] Macedo LG, Smeets RJ, Maher CG, Latimer J, McAuley JH. Graded activity and graded exposure for persistent nonspecific low back pain: a systematic review. Phys Ther. 2010 Jun;90(6):860-79. doi: 10.2522/ptj.20090303. Epub 2010 Apr 15. PMID 20395306
- [Background] Webster F, Perruccio AV, Jenkinson R, Jaglal S, Schemitsch E, Waddell JP, Venkataramanan V, Bytautas J, Davis AM. Understanding why people do or do not engage in activities following total joint replacement: a longitudinal qualitative study. Osteoarthritis Cartilage. 2015 Jun;23(6):860-7. doi: 10.1016/j.joca.2015.02.013. Epub 2015 Feb 21. PMID 25707933
- [Background] Dawson J, Fitzpatrick R, Carr A, Murray D. Questionnaire on the perceptions of patients about total hip replacement. J Bone Joint Surg Br. 1996 Mar;78(2):185-90. PMID 8666621
- [Background] Beard DJ, Harris K, Dawson J, Doll H, Murray DW, Carr AJ, Price AJ. Meaningful changes for the Oxford hip and knee scores after joint replacement surgery. J Clin Epidemiol. 2015 Jan;68(1):73-9. doi: 10.1016/j.jclinepi.2014.08.009. Epub 2014 Oct 31. PMID 25441700
- [Background] Kaplan RS, Anderson SR. Time-driven activity-based costing. Harv Bus Rev. 2004 Nov;82(11):131-8, 150. PMID 15559451
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Husted H. Fast-track hip and knee arthroplasty: clinical and organizational aspects. Acta Orthop Suppl. 2012 Oct;83(346):1-39. doi: 10.3109/17453674.2012.700593. PMID 23205862
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, part I: critical appraisal of existing treatment guidelines and systematic review of current research evidence. Osteoarthritis Cartilage. 2007 Sep;15(9):981-1000. doi: 10.1016/j.joca.2007.06.014. Epub 2007 Aug 27. PMID 17719803
- [Background] Withers TM, Lister S, Sackley C, Clark A, Smith TO. Is there a difference in physical activity levels in patients before and up to one year after unilateral total hip replacement? A systematic review and meta-analysis. Clin Rehabil. 2017 May;31(5):639-650. doi: 10.1177/0269215516673884. Epub 2016 Oct 23. PMID 27773874
- [Background] Jones CA, Martin RS, Westby MD, Beaupre LA. Total joint arthroplasty: practice variation of physiotherapy across the continuum of care in Alberta. BMC Health Serv Res. 2016 Nov 4;16(1):627. doi: 10.1186/s12913-016-1873-9. PMID 27809849